CLINICAL TRIAL: NCT02759107
Title: A Single- and Multiple-Ascending Dose Study in Healthy Subjects to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3298176 and Multiple Doses in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide (LY3298176) in Healthy Participants and Participants With Type 2 Diabetes (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16119; I8F-MC-GPGA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Healthy; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Tirzepatide (Part A) (Experimental): Participants received escalating single doses of either 0.25 milligram (mg) or 0.5mg or 1mg, or 2.5mg or 5mg or 8mg Tirzepatide by subcutaneous injection.
  Interventions: Drug: Tirzepatide
- Placebo (Part A) (Placebo Comparator): Participants received single dose of placebo by subcutaneous injection.
  Interventions: Drug: Placebo
- Tirzepatide (Part B) (Experimental): Participants received fixed doses of either 0.5mg or 1.5mg or 4.5mg Tirzepatide once weekly for four weeks or titrated doses of 5mg, 5mg, 8mg and 10mg Tirzepatide once weekly for four weeks by subcutaneous injection.
  Interventions: Drug: Tirzepatide
- Placebo (Part B) (Placebo Comparator): Participants received placebo once weekly for four weeks by subcutaneous injection.
  Interventions: Drug: Placebo
- Dulaglutide (Part B) (Active Comparator): Participants received 1.5mg Dulaglutide once weekly for four weeks by subcutaneous injection.
  Interventions: Drug: Dulaglutide
- Tirzepatide (Part C) (Experimental): Participants received fixed doses of either 0.5mg or 5mg Tirzepatide once weekly for four weeks or titrated doses of 5mg,5mg,10mg,10mg or 5mg,5mg,10mg,15mg Tirzepatide once weekly for four weeks by subcutaneous injection
  Interventions: Drug: Tirzepatide
- Placebo (Part C) (Placebo Comparator): Participants received placebo once weekly for four weeks by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide (Part A); Tirzepatide (Part B); Tirzepatide (Part C)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)
Drug: Dulaglutide — Administered SC
  Other Names: Trulicity®
  Arms: Dulaglutide (Part B)

SUMMARY:
The main purposes of this study are to determine:

* The safety of tirzepatide and any side effects that might be associated with it.
* How much tirzepatide gets into the bloodstream and how long it takes the body to get rid of it.
* How tirzepatide affects the levels of blood sugar.

This study includes 3 parts (A, B and C). Part A involves a single dose of tirzepatide taken as a subcutaneous (SC) injection just under the skin and will be approximately 10 weeks in duration, including screening. Parts B and C involve 4 doses of tirzepatide taken once weekly (over 4 weeks) as a SC injection just under the skin and is approximately 12-14 weeks in duration, including screening. Each participant will enroll in only one part.

This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (Parts A and B) and participants with T2DM diagnosed at least 1 year before enrollment (Part C)
* Have a screening body mass index (BMI) of greater than 18.5 and less than or equal to 40.0 kilograms per meter squared (kg/m²), inclusive
* Participants with T2DM (Part C only): have T2DM controlled with diet and exercise alone or are stable on a single oral antidiabetic medication (metformin for at least 30 days or sulfonylureas). Participants receiving sulfonylureas may participate only if this treatment is stopped for at least 6 weeks before dosing with study drug

Exclusion Criteria:

* Have known allergies to tirzepatide, glucagon-like peptide (GLP)-1 analogs, or related compounds
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase (greater than 2-fold the upper limit of normal [ULN]) or gastrointestinal (GI) disorder (for example, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (for example, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase (DPP)-IV inhibitors

Participants with T2DM (Part C only)

* Have had more than 1 episode of severe hypoglycemia, as defined by the American Diabetes Association criteria, within 6 months before entry into the study or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms

All Study Participants (Parts B and C only)

* have known allergies to tirzepatide, GLP-1 analogs, or related compounds, or acetaminophen

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Miami Research Associates, South Miami, Florida, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Coskun T, Sloop KW, Loghin C, Alsina-Fernandez J, Urva S, Bokvist KB, Cui X, Briere DA, Cabrera O, Roell WC, Kuchibhotla U, Moyers JS, Benson CT, Gimeno RE, D'Alessio DA, Haupt A. LY3298176, a novel dual GIP and GLP-1 receptor agonist for the treatment of type 2 diabetes mellitus: From discovery to clinical proof of concept. Mol Metab. 2018 Dec;18:3-14. doi: 10.1016/j.molmet.2018.09.009. Epub 2018 Oct 3. PMID 30473097
- See also: Click here for more information about this study:A Study of tirzepatide in Participants With Type 2 Diabetes (T2DM) — https://www.lillytrialguide.com/en-US/studies/type-2-diabetes/GPGA#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Placebo: Participants received placebo by subcutaneous (SC) injection.
- Part A 0.25 mg Tirzepatide: Participants received single dose of 0.25 milligram (mg) Tirzepatide by subcutaneous injection.
- Part A 0.5mg Tirzepatide: Participants received single dose of 0.5mg Tirzepatide by subcutaneous injection.
- Part A 1mg Tirzepatide: Participants received single dose of 1mg Tirzepatide by subcutaneous injection.
- Part A 2.5mg Tirzepatide: Participants received single dose of 2.5mg Tirzepatide by subcutaneous injection.
- Part A 5mg Tirzepatide: Participants received single dose of 5mg Tirzepatide by subcutaneous injection.
- Part A 8mg Tirzepatide: Participants received single dose of 8mg Tirzepatide by subcutaneous injection.
- Part B Placebo; Part C Placebo: Participants received placebo by subcutaneous injection.
- Part B 1.5mg Dulaglutide: Participants received 1.5mg Dulaglutide once weekly for four weeks by subcutaneous injection.
- Part B 0.5mg Tirzepatide; Part C 0.5mg Tirzepatide: Participants received 0.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B 1.5mg Tirzepatide: Participants received 1.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B 4.5mg Tirzepatide: Participants received 4.5mg Tirzepatide once weekly for four weeks by subcutaneous injections.
- Part B 5, 5, 8,10mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 8mg QW followed by 10mg QW.
- Part C 5mg Tirzepatide: Participants received 5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part C 5, 5, 10,10mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 10mg QW followed by 10mg QW.
- Part C 5, 5, 10,15mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 10mg QW followed by 15mg QW.
Period: Overall Study
Arm/Group | Part A Placebo | Part A 0.25 mg Tirzepatide | Part A 0.5mg Tirzepatide | Part A 1mg Tirzepatide | Part A 2.5mg Tirzepatide | Part A 5mg Tirzepatide | Part A 8mg Tirzepatide | Part B Placebo | Part B 1.5mg Dulaglutide | Part B 0.5mg Tirzepatide | Part B 1.5mg Tirzepatide | Part B 4.5mg Tirzepatide | Part B 5, 5, 8,10mg Tirzepatide | Part C Placebo | Part C 0.5mg Tirzepatide | Part C 5mg Tirzepatide | Part C 5, 5, 10,10mg Tirzepatide | Part C 5, 5, 10,15mg Tirzepatide
Started | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 11 | 9 | 9 | 12 | 12
Received at Least One Dose of Study Drug | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 11 | 9 | 9 | 12 | 12
Completed | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 5 | 6 | 6 | 5 | 11 | 9 | 8 | 12 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Not completed — Scheduling Conflict | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Part A 0.25 mg Tirzepatide: Participants received single dose of 0.25mg Tirzepatide by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Part A Placebo | Part A 0.25 mg Tirzepatide | Part A 0.5mg Tirzepatide | Part A 1mg Tirzepatide | Part A 2.5mg Tirzepatide | Part A 5mg Tirzepatide | Part A 8mg Tirzepatide | Part B Placebo | Part B 1.5mg Dulaglutide | Part B 0.5mg Tirzepatide | Part B 1.5mg Tirzepatide | Part B 4.5mg Tirzepatide | Part B 5, 5, 8,10mg Tirzepatide | Part C Placebo | Part C 0.5mg Tirzepatide | Part C 5mg Tirzepatide | Part C 5, 5, 10,10mg Tirzepatide | Part C 5, 5, 10,15mg Tirzepatide | Total
Number analyzed (Participants) | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 11 | 9 | 9 | 12 | 12 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 12 | 4 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 12 | 11 | 133
  >=65 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 4 | 6 | 7 | 2 | 6 | 34
  Male | 14 | 5 | 11 | 4 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 0 | 7 | 7 | 3 | 2 | 10 | 6 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9 | 8 | 7 | 12 | 46
  Not Hispanic or Latino | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 1 | 0 | 1 | 5 | 0 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 13 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 5 | 7 | 1 | 0 | 1 | 5 | 0 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 4
  White | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 9 | 7 | 7 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 14 | 6 | 12 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 1 | 0 | 1 | 5 | 0 | 96
  United States | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9 | 8 | 7 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs)
Description: Number of participants with one or more SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, were reported in the Reported Adverse Events module
Time Frame: Baseline through Day 43 (Part A) and Day 57 (Part B and C)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Tirzepatide (Part A): Participants received escalating doses of either 0.25mg or 0.5mg or 1mg, or 2.5mg or 5mg or 8mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Placebo (Part A); Placebo (Part B); Placebo (Part C): Participants received placebo once weekly for four weeks by subcutaneous injection.
- Tirzepatide (Part B): Participants received escalating doses of either 0.5mg or 1.5mg or 4.5mg or titrated doses of 5mg, 5mg, 8mg and 10mg once weekly for four weeks by subcutaneous injection.
- Tirzepatide (Part C): Participants received either 0.5mg or 5mg or titrated doses of 5mg,5mg,10mg,10mg or 5mg,5mg,10mg,15mg Tirzepatide once weekly for four weeks by subcutaneous injection
Arm/Group | Tirzepatide (Part A) | Placebo (Part A) | Tirzepatide (Part B) | Placebo (Part B) | Dulaglutide (Part B) | Tirzepatide (Part C) | Placebo (Part C)
Number analyzed (Participants) | 42 | 14 | 25 | 4 | 4 | 42 | 11
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide in Part A.
Description: Area under the concentration versus time curve from zero to infinity (AUC [0-∞]) of Tirzepatide in Part A.
Time Frame: Predose, 8hours(h), 24h,48h,72h,96h,120h,168h,336h postdose, day 29, day 43
Population: All randomized participants in part A who received at least one dose of Tirzepatide and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour * nanogram per milliliter (h*ng/mL)
Groups:
- Part A - 0.25mg Tirzepatide: Participants received single dose of 0.25mg Tirzepatide by subcutaneous injection.
- Part A - 0.5mg Tirzepatide: Participants received single dose of 0.5mg Tirzepatide by subcutaneous injection.
- Part A - 1mg Tirzepatide: Participants received single dose of 1mg Tirzepatide by subcutaneous injection.
- Part A - 2.5mg Tirzepatide: Participants received single dose of 2.5mg Tirzepatide by subcutaneous injection.
- Part A - 5mg Tirzepatide; Part A - 8mg Tirzepatide: Participants received single dose of 5mg Tirzepatide by subcutaneous injection.
Arm/Group | Part A - 0.25mg Tirzepatide | Part A - 0.5mg Tirzepatide | Part A - 1mg Tirzepatide | Part A - 2.5mg Tirzepatide | Part A - 5mg Tirzepatide | Part A - 8mg Tirzepatide
Number analyzed (Participants) | 6 | 12 | 5 | 6 | 5 | 7
Hour * nanogram per milliliter (h*ng/mL) | 5760 (22) | 12000 (24) | 22600 (14) | 53200 (36) | 90500 (15) | 169000 (8)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide in Part B
Description: Area under the concentration versus time curve during 1 dosing interval (AUC [0-τ]) of Tirzepatide in Part B. τ equals 168 hours.
Time Frame: Predose, 8hours(h), 24h,48h,72h,168h postdose
Population: All randomized participants in part B who received at least one dose of the Tirzepatide and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour * nanogram per milliliter (h*ng/mL)
Groups:
- Part B - 0.5mg Tirzepatide: Participants received 0.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B - 1.5mg Tirzepatide: Participants received 1.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B - 4.5mg Tirzepatide: Participants received 4.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B - 5, 5, 8,10mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 8mg QW followed by 10mg QW.
Arm/Group | Part B - 0.5mg Tirzepatide | Part B - 1.5mg Tirzepatide | Part B - 4.5mg Tirzepatide | Part B - 5, 5, 8,10mg Tirzepatide
Number analyzed (Participants) | 6 | 6 | 6 | 7
Hour * nanogram per milliliter (h*ng/mL) | 6000 (23) | 16300 (13) | 53300 (19) | 56900 (10)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide in Part C
Description: Area under the concentration versus time curve during 1 dosing interval (AUC [0-τ]) of Tirzepatide in Part C. τ equals 168 hours.
Time Frame: Predose, 8hours(h), 24h,48h,72h,168h postdose
Population: All randomized participants in part C who received at least one dose of Tirzepatide and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour * nanogram per milliliter (h*ng/mL)
Groups:
- Part C - 0.5mg Tirzepatide: Participants received 0.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part C - 5mg Tirzepatide: Participants received 5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part C - 5, 5, 10,10mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 10mg QW followed by 10mg QW.
- Part C - 5, 5, 10,15mg Tirzepatide: Participants received titrated doses of Tirzepatide once a week for four weeks by subcutaneous injection. 5mg QW followed by 5mg QW followed by 10mg QW followed by 15mg QW.
Arm/Group | Part C - 0.5mg Tirzepatide | Part C - 5mg Tirzepatide | Part C - 5, 5, 10,10mg Tirzepatide | Part C - 5, 5, 10,15mg Tirzepatide
Number analyzed (Participants) | 9 | 8 | 12 | 10
Hour * nanogram per milliliter (h*ng/mL) | 4770 (30) | 50500 (20) | 41900 (26) | 37990 (21)

5. Secondary Outcome: Pharmacodynamics (PD): Ratio of AUC of Glucose on Day 2 to Baseline (Part C)
Description: PD: Glucose area under the concentration versus time curve from time 0 to 2 hours (AUC[0-2h]) in Part C. Ratio to Baseline (Day -1) AUC (0-2h).
Time Frame: Pre-glucose dose, 0.5, 1, 1.5, 2 hours post-glucose dose on Day -1 and Day 2
Population: All randomized participants in part C who received at least one dose of Tirzepatide and had evaluable day 2 PD data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part C - 0.5mg Tirzepatide | Part C - 5mg Tirzepatide | Part C - 5, 5, 10,10mg Tirzepatide | Part C - 5, 5, 10,15mg Tirzepatide
Number analyzed (Participants) | 9 | 9 | 12 | 12
ratio | 0.99 [0.79 to 1.11] | 0.72 [0.58 to 0.81] | 0.65 [0.53 to 0.73] | 0.73 [0.59 to 0.81]

6. Secondary Outcome: Pharmacodynamics (PD): Ratio of AUC of Glucose on Day 23 to Baseline (Part C)
Description: as for outcome 5
Time Frame: Pre-glucose dose, 0.5, 1, 1.5, 2 hours post-glucose dose on Day -1 and Day 23
Population: All randomized participants in part C who received at least one dose of Tirzepatide and had evaluable day 23 PD data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part C - 0.5mg Tirzepatide | Part C - 5mg Tirzepatide | Part C - 5, 5, 10,10mg Tirzepatide | Part C - 5, 5, 10,15mg Tirzepatide
Number analyzed (Participants) | 9 | 7 | 12 | 11
ratio | 0.96 [0.83 to 1.16] | 0.61 [0.52 to 0.75] | 0.58 [0.51 to 0.70] | 0.57 [0.50 to 0.69]

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 57 days)
Description: All randomized participants who received at least 1 dose of the study drug.
Groups:
- Part A - Placebo: Participants received placebo by subcutaneous (SC) injection.
- Part A - 0.25mg Tirzepatide: Participants received 0.25mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part A - 0.5mg Tirzepatide; Part B - 0.5mg Tirzepatide; Part C - 0.5mg Tirzepatide: Participants received 0.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part A - 1mg Tirzepatide: Participants received 1mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part A - 2.5mg Tirzepatide: Participants received 2.5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part A - 5mg Tirzepatide; Part C - 5mg Tirzepatide: Participants received 5mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part A - 8mg Tirzepatide: Participants received 8mg Tirzepatide once weekly for four weeks by subcutaneous injection.
- Part B - Placebo; Part C - Placebo: Participants received placebo by subcutaneous injection.
- Part B - 1.5mg Dulaglutide: Participants received 1.5mg Dulaglutide once weekly for four weeks by subcutaneous injection.
- Part B - 4.5mg Tirzepatide: Participants received 4.5mg Tirzepatide once weekly for four weeks by subcutaneous injections.
Arm/Group | Part A - Placebo | Part A - 0.25mg Tirzepatide | Part A - 0.5mg Tirzepatide | Part A - 1mg Tirzepatide | Part A - 2.5mg Tirzepatide | Part A - 5mg Tirzepatide | Part A - 8mg Tirzepatide | Part B - Placebo | Part B - 1.5mg Dulaglutide | Part B - 0.5mg Tirzepatide | Part B - 1.5mg Tirzepatide | Part B - 4.5mg Tirzepatide | Part B - 5, 5, 8,10mg Tirzepatide | Part C - Placebo | Part C - 0.5mg Tirzepatide | Part C - 5mg Tirzepatide | Part C - 5, 5, 10,10mg Tirzepatide | Part C - 5, 5, 10,15mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/12 | 0/5 | 0/6 | 0/6 | 0/7 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/7 | 0/11 | 0/9 | 0/9 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/12 | 0/5 | 0/6 | 0/6 | 0/7 | 0/4 | 1/4 | 0/6 | 0/6 | 0/6 | 0/7 | 0/11 | 0/9 | 0/9 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/14 | 4/6 | 10/12 | 3/5 | 2/6 | 6/6 | 7/7 | 3/4 | 3/4 | 6/6 | 5/6 | 6/6 | 6/7 | 3/11 | 5/9 | 7/9 | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Placebo (N=14) | Part A - 0.25mg Tirzepatide (N=6) | Part A - 0.5mg Tirzepatide (N=12) | Part A - 1mg Tirzepatide (N=5) | Part A - 2.5mg Tirzepatide (N=6) | Part A - 5mg Tirzepatide (N=6) | Part A - 8mg Tirzepatide (N=7) | Part B - Placebo (N=4) | Part B - 1.5mg Dulaglutide (N=4) | Part B - 0.5mg Tirzepatide (N=6) | Part B - 1.5mg Tirzepatide (N=6) | Part B - 4.5mg Tirzepatide (N=6) | Part B - 5, 5, 8,10mg Tirzepatide (N=7) | Part C - Placebo (N=11) | Part C - 0.5mg Tirzepatide (N=9) | Part C - 5mg Tirzepatide (N=9) | Part C - 5, 5, 10,10mg Tirzepatide (N=12) | Part C - 5, 5, 10,15mg Tirzepatide (N=12)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A - Placebo (N=14) | Part A - 0.25mg Tirzepatide (N=6) | Part A - 0.5mg Tirzepatide (N=12) | Part A - 1mg Tirzepatide (N=5) | Part A - 2.5mg Tirzepatide (N=6) | Part A - 5mg Tirzepatide (N=6) | Part A - 8mg Tirzepatide (N=7) | Part B - Placebo (N=4) | Part B - 1.5mg Dulaglutide (N=4) | Part B - 0.5mg Tirzepatide (N=6) | Part B - 1.5mg Tirzepatide (N=6) | Part B - 4.5mg Tirzepatide (N=6) | Part B - 5, 5, 8,10mg Tirzepatide (N=7) | Part C - Placebo (N=11) | Part C - 0.5mg Tirzepatide (N=9) | Part C - 5mg Tirzepatide (N=9) | Part C - 5, 5, 10,10mg Tirzepatide (N=12) | Part C - 5, 5, 10,15mg Tirzepatide (N=12)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (7) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (13) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (29) | 0 (0) | 1 (3) | 0 (0) | 1 (4) | 9 (33)
Administration site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (9) | 4 (9) | 1 (1) | 2 (2) | 6 (7) | 5 (11) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food aversion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/4 (0) | 1/6 (1) | 0/7 (0) | 0/2 (0) | 0/6 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT02759107/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02759107/SAP_001.pdf